CLINICAL TRIAL: NCT02532023
Title: The Combined Effects of omega3 Fatty Acids and Curcumin Supplementation on Gene Expression and Serum Levels of Some Inflammatory and Endothelial Factors in Migraine Patients
Brief Title: The Combined Effects of omega3 Fatty Acids and Curcumin Supplementation on Inflammatory and Endothelial Factors in Migraine Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 28825
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Migraine
Keywords: omega 3 fatty acid; curcumin; COX-2; iNOs; VCAM-1; ICAM-1; IL-1β; IL-6; TNF-α; hsCRP; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Fatty Acids, Omega-3; Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- omega 3 fatty acid supplementation (Active Comparator): patients with migraine receive 2 capsules 1000 mg omega3, 2 times a day, for 2 months.
  Interventions: Dietary Supplement: omega 3 fatty acid
- curcumin supplementation (Active Comparator): patients with migraine receive 2 capsules 1000 mg curcumin, 2 times a day, for 2 months.
  Interventions: Dietary Supplement: curcumin
- omega 3 fatty acid Placebo (Placebo Comparator): patients with migraine receive 2 capsules of omega 3 fatty acid placebo for 2 months.
  Interventions: Dietary Supplement: omega 3 fatty acid placebo
- curcumin placebo (Placebo Comparator): patients with migraine receive 2 capsules of curcumin placebo for 2 months.
  Interventions: Dietary Supplement: curcumin placebo

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acid — omega 3 fatty acid supplement, 2× 1000 mg softgel daily (1800 mg EPA+DHA per day), 2 times a day, for 2 months
  Other Names: n-3 PUFA; n-3 Fatty Acid
  Arms: omega 3 fatty acid supplementation
Dietary Supplement: curcumin — curcumin supplement, 2× 500 mg softgel daily (1000 mg curcumin per day), 2 times a day, for 2 months
  Arms: curcumin supplementation
Dietary Supplement: omega 3 fatty acid placebo — omega 3 fatty acid placebo softgel (Containing 2 g edible paraffin oil), 2× 1000 mg softgel daily (2 g per day), 2 times a day, for 2 months
  Arms: omega 3 fatty acid Placebo
Dietary Supplement: curcumin placebo — curcumin placebo softgel (Containing 1 g starch powder), 2× 500 mg softgel daily (1 g per day), 2 times a day, for 2 months
  Arms: curcumin placebo

SUMMARY:
The aim of this study is to determine the effects of omega 3 fatty acid, curcumin and their combination or placebo for 2 months on the gene expression of COX-2, iNOS, TNF-α, IL-1β, IL-6, VCAM-1 and ICAM-1 in the peripheral blood mononuclear cell (PBMC) and serum levels of COX-2, iNOS, TNF-α, IL-1β, IL-6, VCAM-1, ICAM-1 and hsCRP of migraine patients.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of omega 3 fatty acid, curcumin and their combination or placebo for 2 months on the gene expression of cyclooxygenase-2 (COX-2), inducible nitric oxide synthase (iNOS), Tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β), interleukin-6 (IL-6), vascular cell adhesion molecule-1 (VCAM-1) and intercellular adhesion molecule-1 (ICAM-1) in the peripheral blood mononuclear cell (PBMC) and serum levels of COX-2, iNOS, TNF-α, IL-1β, IL-6, VCAM-1, ICAM-1 and high-sensitivity C-reactive protein (hsCRP) of migraine patients.

In this randomized, double-blind clinical trial, placebo-controlled study, 80 women and men with migraine are enrolled from the Iranian Center of Neurological Research. At the start of study, all participants will sign informed consent and complete a general information form. 24-hour food recall for 3 days will be taken from the patients at the beginning and the end of the study. Selected samples by using stratified randomization method based on sex, gender and body mass index (BMI) are classified into 4 groups: 1) receiving omega 3 fatty acid supplement and curcumin supplement 2) receiving omega 3 fatty acid supplement and curcumin placebo 3) receiving curcumin supplement and omega 3 fatty acid placebo 4) receiving omega 3 fatty acid placebo and curcumin placebo.

The omega 3 fatty acid supplement group will receive 1200 mg Eicosapentaenoic acid (EPA) and 600 mg Docosahexaenoic acid (DHA) totally 1800 mg daily for 2 months. The curcumin supplement group will receive 1000 mg curcumin daily for 2 months. The omega 3 fatty acid placebo group will also receive placebo containing 1800 mg edible paraffin oil and curcumin placebo group will receive 1000 mg starch powder both similar in terms of color, shape and size. participants are advised to maintain their diet, level of physical activity and medication dose during the study. Blood samples will be collected after anthropometric parameter measuring then target biochemical parameters, gene expression and serum levels and physical activity will be measured before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* migraine patients 20- 50 years old
* body mass index more than 18.5
* avoidance of dietary supplements, vitamins and herbal products at least 4-6 weeks before and throughout the intervention
* willingness to participation

Exclusion Criteria:

* sensitivity to omega 3 fatty acid and curcumin
* pregnancy and lactation
* sever change in regular diet and life style
* change in type and dosage of regular medication (s)
* inflammatory disease which need take anti inflammatory drugs over than 2 weeks

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
headache attack | Change frome baseline at 2 months

SECONDARY OUTCOMES:
serum COX-2 | Change frome baseline at 2 months
serum iNOs | Change frome baseline at 2 months
serum VCAM-1 | Change frome baseline at 2 months
serum ICAM-1 | Change frome baseline at 2 months
serum TNF-α | Change frome baseline at 2 months
serum IL-1β | Change frome baseline at 2 months
serum IL-6 | Change frome baseline at 2 months
serum hsCRP | Change frome baseline at 2 months
headache duration | Change frome baseline at 2 months
headache severity | Change frome baseline at 2 months
COX-2 gene expression | Change frome baseline at 2 months
iNOs gene expression | Change frome baseline at 2 months
VCAM-1 gene expression | Change frome baseline at 2 months
ICAM-1 gene expression | Change frome baseline at 2 months
TNF-α gene expression | Change frome baseline at 2 months
IL-1β gene expression | Change frome baseline at 2 months
IL-6 gene expression | Change frome baseline at 2 months

REFERENCES:
- [Derived] Djalali M, Talebi S, Djalali E, Abdolahi M, Travica N, Djalali M. The effect of omega-3 fatty acids supplementation on inflammatory biomarkers in subjects with migraine: a randomized, double-blind, placebo-controlled trial. Immunopharmacol Immunotoxicol. 2023 Oct;45(5):565-570. doi: 10.1080/08923973.2023.2196600. Epub 2023 Apr 26. PMID 37126739
- [Derived] Abdolahi M, Karimi E, Sarraf P, Tafakhori A, Siri G, Salehinia F, Sedighiyan M, Asanjarani B, Badeli M, Abdollahi H, Yoosefi N, Yousefi A, Rad AS, Djalali M. The omega-3 and Nano-curcumin effects on vascular cell adhesion molecule (VCAM) in episodic migraine patients: a randomized clinical trial. BMC Res Notes. 2021 Jul 23;14(1):283. doi: 10.1186/s13104-021-05700-x. PMID 34301320
- [Derived] Abdolahi M, Sarraf P, Javanbakht MH, Honarvar NM, Hatami M, Soveyd N, Tafakhori A, Sedighiyan M, Djalali M, Jafarieh A, Masoudian Y, Djalali M. A Novel Combination of omega-3 Fatty Acids and Nano-Curcumin Modulates Interleukin-6 Gene Expression and High Sensitivity C-reactive Protein Serum Levels in Patients with Migraine: A Randomized Clinical Trial Study. CNS Neurol Disord Drug Targets. 2018;17(6):430-438. doi: 10.2174/1871527317666180625101643. PMID 29938621